CLINICAL TRIAL: NCT03407833
Title: Physiologic and Functional Adaptations of Insulin Sensitive Tissues After Bariatric Surgery
Brief Title: Physiologic and Functional Adaptations of Insulin Sensitive Tissues
Status: Enrolling by invitation | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Charles R. Flynn, Principal Investigator, Vanderbilt University Medical Center
Other Study IDs: 171845
Record Dates: First submitted 2018-01-04; First posted 2018-01-23 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Diabetes; Insulin Resistance; Obesity; Bariatric Surgery Candidate; Roux-en-y Gastric Bypass; Liver Diseases
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance; Obesity; Liver Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsy tissue specimens will be stored in RNAlater© and will be used to measure mRNA expression profiles. Blood and fecal samples will also be obtained and stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Obese, surgery: Obese subjects recruited from the Center for Surgical Weight loss who are undergoing weight loss surgery as part of their standard of care. Tissue biopsies, blood, and fecal swabs will be collected at surgical visits.
  Interventions: Other: Surgical biopsy; Other: Mixed-meal tolerance test
- Obese, nonsurgery: Obese subjects recruited from the Vanderbilt Endoscopy Clinic who are undergoing upper endoscopy or colonoscopy as part of their standard of care. Tissue biopsies, blood, and fecal swabs will be collected at day of procedure.
  Interventions: Other: Endoscopy biopsy
- Lean control: Lean control subjects recruited from the Vanderbilt Endoscopy Clinic who are undergoing upper endoscopy or colonoscopy as part of their standard of care. Tissue biopsies, blood, and fecal swabs will be collected at day of procedure.
  Interventions: Other: Endoscopy biopsy
- Liver transplant: Lean or obese subjects who are undergoing liver transplantation as part of their standard of care. Excised liver tissue will be collected the day of procedure.
  Interventions: Other: Excised Liver Tissue Sampling

INTERVENTIONS:
Other: Endoscopy biopsy — Tissue samples will be collected from the jejunum, duodenum, and colon during the subject's standard of care procedure.
  Groups: Lean control; Obese, nonsurgery
Other: Surgical biopsy — Biopsy of the liver is standard of care for diagnosing NAFLD. Biopsy of omentum, skeletal muscle and subcutaneous adipose (the latter two tissues taken at the site of trocar placement) will be collected intraoperatively at the time of Roux-en-Y gastric bypass (RYGB) or vertical sleeve gastrectomy (VSG).
  Groups: Obese, surgery
Other: Mixed-meal tolerance test — The mixed meal tolerance test (MMTT) shows how much insulin your body is making after drinking a liquid meal beverage that contains fats, protein and carbohydrates (sugar). Glucose, C-peptide, free fatty acids, triglycerides, incretins, pancreatic polypertide, bile aceis, and fatty acid amides can also be measured. A total of 9 tablespoons of blood is taken over a 255 minute period.
  Groups: Obese, surgery
Other: Excised Liver Tissue Sampling — Tissue will be collected from the excised liver for research after the diseased liver has been removed as part of the standard of care procedure.
  Groups: Liver transplant

SUMMARY:
The long-term goal is to understand the mechanisms of intestinal nutrient sensing and signal relays to insulin sensitive tissues (adipose, skeletal muscle, liver) in humans. The investigators hypothesize that human tissue biopsies (from obese surgery and non-surgery subjects as well as lean controls) can be used to understand the molecular mechanisms underlying intestinal nutrient sensing and signal relay in humans. The investigator will obtain tissue specimens from patients during scheduled upper endoscopies, colonoscopies and scheduled metabolic and bariatric surgeries or liver transplantation. A blood sample (4mL) will be obtained concurrent with these procedures. From metabolic and bariatric surgery subjects blood and tissues (liver, adipose, small intestine, omentum, skeletal muscle) can be collected at the time of surgery. From liver transplantation patients, excised liver tissue will be collected. Stool can be obtained preoperatively and at various time points after surgery. Some bariatric surgery subjects will participate in a mixed-meal tolerance test at their pre-operative visit and several post-operative visits to compare the whole-body metabolic alterations following bariatric procedures.

DETAILED DESCRIPTION:
Upper endoscopy (subset)

* Intestinal biopsies will be obtained during scheduled upper endoscopy from the mid-duodenum and/or proximal jejunum. In the case that a patient requires an upper endoscopy after metabolic and bariatric surgery, biopsies will be obtained from the mid-jejunum.
* Blood will be collected from an IV placed in the arm used for administering anesthesia required for the indicated procedure.

Colonoscopy (subset)

* Biopsies of the colon will be obtained during scheduled colonoscopy.
* Blood will be collected from an IV placed in the arm used for administering anesthesia required for the indicated procedure.

Metabolic and bariatric surgery (subset)

* During the metabolic and bariatric surgical procedures, biopsy of the jejunum, liver and omentum (visceral adipose) may be obtained. Biopsies of skeletal muscle and subcutaneous adipose will be taken at the sites of trocar placement for laparotomy.
* Blood will be collected from an IV placed in the arm used for administering anesthesia required for the indicated procedure.
* Feces will be self-collected by the patient using a provided culture swab specimen container or FOB card.

Liver transplantation (subset)

• Tissue will be collected from excised disease liver

ELIGIBILITY:
Inclusion Criteria:

- Scheduled for upper endoscopy, colonoscopy or metabolic and bariatric surgery, or liver transplantation at Vanderbilt University Medical Center.

Additional inclusion criteria for individuals scheduled for metabolic and bariatric surgery: Obese, ≥ 40 kg/m2 or ≥ 35 kg/m2 + one comorbidity (type 2 diabetes [fasting blood glucose ≥ 120 mg/dL; HbA1C ≥ 6.5%]; fatty liver disease, hypertension, cardiovascular disease, hyperlipidemia)

Additional inclusion criteria for individuals scheduled for liver transplantation: diagnosis of nonalcoholic liver disease or nonalcoholic steatohepatitis

Exclusion Criteria:

* Known history of intestinal diseases including, but not limited to, inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease) and celiac sprue.
* Smoking >7 cigarettes per day
* Malabsorptive syndromes
* Pregnant or breastfeeding

Additional exclusion criteria for patients undergoing endoscopy/colonoscopy:

* Recent history of malignancy (<5 years ago)
* Previous lap band surgery
* Established renal disease

Additional exclusion criteria for patients undergoing bariatric surgery:

* Previous lap band, sleeve gastrectomy, or gastric bypass surgery
* Recent history of malignancy (< 5 years ago)
* Established organ dysfunction

Additional exclusion criteria for patients undergoing liver transplantation:

* Previous lap band, sleeve gastrectomy, or gastric bypass surgery
* Alpha 1 anti-trypsin disease, Wilson's disease, viral hepatitis, alcoholic liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese or lean subjects seen in the Vanderbilt Endoscopy Clinic, obese subjects planning surgery at the Center for Surgical Weight Loss, or obese or lean subjects planning liver transplantation surgery will be approached by research staff to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-02-13 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Ability to establish organoid cultures | 12 months
  Measure percent success rate of making organoid cultures from tissue biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Charles Flynn, Ph.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No